CLINICAL TRIAL: NCT04101084
Title: Rocking Chair Therapy: A Non Pharmacological Intervention in Elderly With Dementia, Its Effects in Agitation, Pharmacological Restraint Use, and Pain
Brief Title: Rocking Chair Therapy in Elderly With Dementia: Its Effects on Agitation
Acronym: Rocking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-AOIP-03
Record Dates: First submitted 2019-08-08; First posted 2019-09-24 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: to evaluate the effect of the rocking chair therapy in agitation for home care residents with dementia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rocking chair therapy (Experimental): Rocking sessions in a safe rocking chair for 2 hours daily for six weeks
  Interventions: Other: Therapy

INTERVENTIONS:
Other: Therapy — Rocking sessions in a safe rocking chair for 2 hours daily for six weeks

SUMMARY:
Patients with dementia exhibit a wide range of behavioral symptoms which include mood disturbances (e.g depression, anxiety), behavior and activity disturbances (e.g agitation, aggression, wandering) and psychotic symptoms (e.g hallucinations and delusions). Behavioral disturbances are a major source of caregiver burden and an important contributor to the decision to admit AD patients to institutionalized long-term care.

Among the innovative approaches, rocking chair therapy has been introduced as a potential means for reducing agitation in elderly with dementia. Only few studies evaluated the effect of this therapy on the behavioral symptoms in elderly with cognitive impairment. The results were promising, but not sufficiently significant.

We propose to perform this study having as a main goal to evaluate the effect of the rocking chair therapy in agitation for home care residents with dementia. The secondary aim of the study will be the evaluation of psychoactive drugs use as well as pain killers. Cohen Mansfield agitation inventory will be employed for the pre- and post-therapy evaluation.

Included subjects will be installed in groups of five, rocking chairs will be placed away from other residents in a semicircle in a corner of the dayroom. The therapy sessions will be held every afternoon, for two hours, under the supervision of the unit psychologist and a master's degree psychology student. During the daily session, each resident should be encouraged to actively rock to reach the goal of 60 minutes of rocking accumulated per day. The total duration of the therapy period will be 6 weeks. The use of pharmacological restraint (neuroleptics, anxiolytics) and pain killers will be evaluated before, during and after the six weeks therapy.

The expected outcome is a reduction of agitation among elderly with dementia, as well as a reduction in the use of pharmacological restraint and pain killers.

ELIGIBILITY:
Inclusion Criteria:

* resident of the EHPAD / LTC for at least 10 weeks
* subject with cognitive impairment (MMSE <24) documented according to DSM-5 criteria
* with chronic behavioral disorders such as agitation
* stable from a medical point of view
* without restraint when not in bed
* ability to touch the floor with the toes while sitting in the rocking chair
* ability to sit securely in the rocking chair
* ability to tolerate rocking chair
* Ability to maintain active rocking for at least 5 minutes over a 30-minute period during the three pre-treatment trials
* obligation for all patients to be affiliated to a social security scheme
* signing of the informed consent by the patient and / or his legal representative

Exclusion Criteria:

* Motor deficiency (example: after-effects of stroke ...) not allowing a secure installation in the chair or preventing an active rocking
* ATCC with vestibular involvement that may lead to vertiginous seizures during rocking
* Aging psychiatric pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2024-04-18 (Estimated)

PRIMARY OUTCOMES:
Change of agitation | At 6 weeks
  Change from Baseline agitation at 6 weeks. The agitation will be evaluated using Cohen Mnasfiled agitation inventory a week before therapy, and the week after.

CONTACTS AND LOCATIONS:
Overall Officials: ZAAFRANE Malek, Ph, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Gérontology, Nice, Alpes-Maritime, France

IPD SHARING:
Plan to Share IPD: No